CLINICAL TRIAL: NCT01766778
Title: A Local Phase IV, Multicenter, Open-label Study to Evaluate Early add-on Vildagliptin in Patients With Type 2 Diabetes Inadequately Controlled by Metformin
Brief Title: Early add-on Vildagliptin in Patients With Type 2 Diabetes Inadequately Controlled by Metformin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLAF237AHK01
Record Dates: First submitted 2013-01-09; First posted 2013-01-11 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Type-2 Diabetes Mellitus
Keywords: type-2 diabetes mellitus, inadequately controlled Metformin
MeSH Terms: interventions — 1-(((3-hydroxy-1-adamantyl)amino)acetyl)-2-cyanopyrrolidine; Vildagliptin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LAF237 (vildagliptin) 50mg once daily (QD) (Active Comparator): Vildagliptin 50mg QD plus stabilized or maximum tolerated dose of Metformin
  Interventions: Drug: LAF237 (vildagliptin); Drug: Metformin
- LAF237 (vildagliptin) 50mg twice daily (BID) (Active Comparator): Vildagliptin 50mg BID plus stabilized or maximum tolerated dose of Metformin
  Interventions: Drug: LAF237 (vildagliptin); Drug: Metformin

INTERVENTIONS:
Drug: LAF237 (vildagliptin) — Vildagliptin 50mg capsule
  Other Names: LAF237
Drug: Metformin — Metformin maximum tolerance dose

SUMMARY:
The purpose of this study was to observe change of HbA1c over time from baseline to month 12. The ultimate goal of this study was to provide a local reference value to the physicians & patients in the future when they consider initiating Vildagliptin and taking balance between efficacy, compliance, risk factors, convenience and medication cost.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female in age ≥18 at Visit 1
2. Type 2 diabetes mellitus (T2DM) patients on their maximum tolerated dose of Metformin for more than 3 months
3. HbA1c (glycosylated hemoglobin) at Visit 1 greater than 7.0%
4. With nearest documented record of HbA1c before Visit 1 greater than 7.0% after patient reached his/her maximum tolerated dose of Metformin

Key Exclusion Criteria:

1. Patients with hepatic impairment, including patients with a pre-treatment alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 X the upper limit of normal at Visit 1
2. Patients with moderate or severe renal impairment or end-stage-renal-disease (ESRD) on haemodialysis at the time of enrolment
3. Patients with hereditary problems of galactose intolerance, the Lapp lactose deficiency or glucose-galactose malabsorption
4. Pregnant women or breastfeeding women at the time of enrolment
5. Use of insulin or other oral anti-diabetic drug (OAD) apart from Metformin in the past for T2DM treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2013-05-13 (Actual); Primary Completion 2015-10-22 (Actual); Study Completion 2015-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Hong Kong (4):
  - Novartis Investigative Site, Hong Kong, Hong Kong
  - Novartis Investigative Site, Tuenmen, Hong Kong
  - Novartis Investigative Site, Hong Kong
  - Novartis Investigative Site, Hong Kong SAR

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was 117 patients randomized and received either Vildagliptin 50mg QD or 50 mg BID.
Period: Overall Study
Arm/Group | LAF237 (Vildagliptin) 50mg Once Daily (QD) | LAF237 (Vildagliptin) 50mg Twice Daily (BID)
Started | 56 (Intent to treat population) | 61
Completed | 51 | 57
Not Completed | 5 | 4
Not completed — Adverse Event | 4 | 4
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) included all randomized patients who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | LAF237 (Vildagliptin) 50mg Once Daily (QD) | LAF237 (Vildagliptin) 50mg Twice Daily (BID) | Total
Number analyzed (Participants) | 56 | 61 | 117
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58 (10.3) | 59 (10.0) | 58 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 31 | 57
  Male | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change of Glycosylated Hemoglobin A1c (HbA1c) From Baseline to Month 12
Description: HbA1c is an integrated measure of average glucose concentration in plasma in the last 2-3 months. Blood samples were collected to analyze HbA1c
Time Frame: Baseline, Month 12 (weeK 52)
Population: Intent to treat (ITT) analysis set included all randomized patients who received at least one dose of study medication. Patients with both baseline and 12 month data were included in this analysis
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | LAF237 (Vildagliptin) 50mg Once Daily (QD) | LAF237 (Vildagliptin) 50mg Twice Daily (BID)
Number analyzed (Participants) | 49 | 50
percentage of Glycosylated Hemoglobin | -0.8 (1.01) | -1.0 (1.24)

2. Secondary Outcome: Change of Glycosylated Hemoglobin A1c (HbA1c) From Baseline to Month 3, 6, 9 and 12 (Based on MMRM Analysis)
Description: HbA1c is an integrated measure of average glucose concentration in plasma in the last 2-3 months. Blood samples were collected to analyze HbA1c. Mixed Model of Repeated Measures (MMRM) was used to analyze this outcome. For the MMRM analysis, the model includes terms for treatment, period, treatment-by-period interaction and baseline value, and further adjusted by age, pre-existing hypertension and microvascular and macrovascular complications for diabetes mellitus. The variables selected for baseline adjustment were based on the lowest AIC.
Time Frame: Baseline, Month 3, 6, 9 and 12
Population: Intent to treat (ITT) analysis set included all randomized patients who received at least one dose of study medication. .
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | LAF237 (Vildagliptin) 50mg Once Daily (QD) | LAF237 (Vildagliptin) 50mg Twice Daily (BID)
Number analyzed (Participants) | 56 | 61
percentage of Glycosylated Hemoglobin
  3 month from baseline | -0.6 (0.11) | -0.9 (0.10)
  6 month from baseline | -0.7 (0.13) | -0.9 (0.12)
  9 month from baseline | -0.7 (0.13) | -0.7 (0.13)
  12 month from baseline | -0.6 (0.15) | -0.6 (0.15)

3. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Month 3, 6, 9 and 12 (Based on MMRM Analysis)
Description: Blood samples were collected to analyze fasting plasma glucose. Mixed Model of Repeated Measures (MMRM) was used to analyze this outcome. For the MMRM analysis, the model included terms for treatment, period, treatment-by-period interaction and baseline value, and further adjusted by pre-existing hypertension. The variable selected for baseline adjustment was based on the lowest AIC.
Time Frame: Baseline, Month 3, 6, 9 and 12
Population: Intent to treat (ITT) analysis set included all randomized patients who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | LAF237 (Vildagliptin) 50mg Once Daily (QD) | LAF237 (Vildagliptin) 50mg Twice Daily (BID)
Number analyzed (Participants) | 56 | 61
mmol/L
  3 month from baseline | -0.9 (0.18) | -1.3 (0.16)
  6 month from baseline | -1.2 (0.18) | -0.9 (0.17)
  9 month from baseline | -1.1 (0.17) | -1.0 (0.16)
  12 month from baseline | -0.9 (0.20) | -0.8 (0.20)

4. Secondary Outcome: Percentage of Patients Achieving Good Glycemic Control
Description: Blood samples were collected to analyze HbA1c. Good glycemic control is defined as patient achieving Hb1Ac < 7.0%. Percentage of patients who achieved HbA1c less than 7.0% at month 3, 6, 9 and 12 were reported for this endpoint.
Time Frame: Month 3, 6, 9, 12
Population: Intent to treat (ITT) analysis set included all randomized patients who received at least one dose of study medication. 'n' indicates patients with HbA1c data in that time point.
Measure: Number; unit: Percentage of patients
Arm/Group | LAF237 (Vildagliptin) 50mg Once Daily (QD) | LAF237 (Vildagliptin) 50mg Twice Daily (BID)
Number analyzed (Participants) | 56 | 61
Percentage of patients
  At Month 3: number analyzed (Participants) | 51 | 59
  At Month 3 | 33.3 | 47.5
  At Month 6: number analyzed (Participants) | 51 | 57
  At Month 6 | 39.2 | 45.6
  At Month 9: number analyzed (Participants) | 51 | 57
  At Month 9 | 45.1 | 47.4
  At Month 12: number analyzed (Participants) | 49 | 50
  At Month 12 | 49.0 | 40.0

5. Secondary Outcome: Percentage of Overall Drug Compliance in 12 Months
Description: The overall drug compliance (%) = (Observed Consumption / Expected Consumption) x 100% Where (Observed Consumption / Expected Consumption) = [1- (Number of missing tablets from all visits/(sum of Allocated Daily Dosage (in tablets) from all visits × No. of Days between the Date Dispensed and the Date Returned))]
Time Frame: Month 12
Population: Intent to treat (ITT) analysis set included all randomized patients who received at least one dose of study medication. Patients who had reported dosing compliance were included in this analysis.
Measure: Mean (Standard Deviation); unit: Percentage of overall drug compliance
Arm/Group | LAF237 (Vildagliptin) 50mg Once Daily (QD) | LAF237 (Vildagliptin) 50mg Twice Daily (BID)
Number analyzed (Participants) | 21 | 21
Percentage of overall drug compliance | 96.90 (5.682) | 97.48 (6.277)

6. Secondary Outcome: Number of Patients With Adverse Events, Serious Adverse Events and Death as an Assessment of Overall Safety and Tolerability
Description: This analysis reported percentage patients with adverse events and patient discontinued from the study due to adverse events. Aslo, percentage of patients with serious adverse events and death was reported.
Time Frame: Month 12
Population: Intent to treat (ITT) analysis set included all randomized patients who received at least one dose of study medication.
Measure: Number; unit: Patients
Arm/Group | LAF237 (Vildagliptin) 50mg Once Daily (QD) | LAF237 (Vildagliptin) 50mg Twice Daily (BID)
Number analyzed (Participants) | 56 | 61
Patients
  Any adverse events | 15 | 14
  Serious adverse events | 2 | 2
  Death | 0 | 0
  Patients discontinued due to any AE/SAE | 4 | 4

ADVERSE EVENTS:
Arm/Group | LAF237 (Vildagliptin) 50mg Once Daily (QD) | LAF237 (Vildagliptin) 50mg Twice Daily (BID)
Serious Adverse Events (participants affected / at risk) | 2/56 | 2/61
Other Adverse Events (participants affected / at risk) | 14/56 | 7/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LAF237 (Vildagliptin) 50mg Once Daily (QD) (N=56) | LAF237 (Vildagliptin) 50mg Twice Daily (BID) (N=61)
Duodenitis (Gastrointestinal disorders) | 1 | 0
Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
stone impairation over proximal urethra (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LAF237 (Vildagliptin) 50mg Once Daily (QD) (N=56) | LAF237 (Vildagliptin) 50mg Twice Daily (BID) (N=61)
Tinea (Infections and infestations) | 0 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 8 | 2
Elevated liver function test (Investigations) | 2 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 2
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0
Dizziness (Nervous system disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Eczema (Skin and subcutaneous tissue disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.